CLINICAL TRIAL: NCT07060300
Title: Comprehensive Assessment of Reactions to Pharmacogenetics in Complex Care Patients
Acronym: CAREPICC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Sonya Tang Girdwood, Associate Professor of Pediatrics, Children's Hospital Medical Center, Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025-0139
Record Dates: First submitted 2025-06-03; First posted 2025-07-11 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Pediatric Medical Complexity Based on PMCA Score of 3
Keywords: Medical Compexity; Pharmacogenetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Accept Pharmacogenetic Testing (Experimental): Caregivers who agree to receive Pharmacogenetic testing for their child
  Interventions: Other: Agree to Pharmacogenetic Testing

INTERVENTIONS:
Other: Agree to Pharmacogenetic Testing — Caregivers agree to receive pharmacogenetic testing for their child.

SUMMARY:
The goal of this clinical trial is to determine the feasibility and acceptability of Pharmacogenetic Testing, and the attitudes towards the same in caregivers of complex care patients in Cincinnati, OH. The main question[s] it aims to answer are:

1. With financial and access barriers removed, do caregivers of complex care patients agree to receive Pharmacogenetic testing for their children?
2. With financial and access barriers removed, what are some remaining barriers to implementation of pharmacogenetics testing?
3. What are the prevailing attitudes towards Pharmacogenetic testing in the complex care population?

Participants will be offered pharmacogenetic testing for their child free of charge, and will be asked to fill out a voluntary survey. Certain caregivers of complex care patients may be asked if they want to participate in a short semi-structured interview.

DETAILED DESCRIPTION:
Through this research, the investigators expect to have successfully provided pharmacogenetic testing to a large cohort of patients in Cincinnati Children's Complex Care Clinic, allowing for an improved understanding of how to provide pharmacogenetic testing in children with medical complexity (feasibility) and of caregiver attitudes about pharmacogenetic testing for their children (acceptability). The knowledge gained from this study will be used to inform future program implementations in children with medical complexity (CMC) populations. Successfully tested patients will also provide for future studies to measure the effectiveness of pharmacogenetic testing in this population, as well as prescriber behavior when provided pharmacogenetic testing results.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who score a 3 on the Pediatric Medical Complexity Algorithm
2. Patients whose primary care providers are those at the Cincinnati Children's Complex Care Clinic

   1. Patients attending the Cincinnati Children's Hospital Complex Care Clinic for well child visit
   2. Patients attending the Cincinnati Children's Hospital Complex Care Clinic for chronic care management visits
   3. Legal Guardian is present at time of clinical visit

Exclusion Criteria:

* Patients attending the Complex Care Clinic for acute illness.
* Patients who have previously received Pharmacogenetic Testing.
* Patients deemed ineligible for approach by the clinical team.
* Patients who are wards of the state.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Caregivers of Medically Complex Patients who accept the offer of Free Clinical Pharmacogenetic Testing | Day 1
  What portion of caregivers accept pharmacogenetic testing for their children when the barriers of access and financial burden are removed

SECONDARY OUTCOMES:
Barriers to acceptance of Pharmacogenetic testing | 6 months
  Barriers will be elicited through semi-structured interviews on consenting caregivers. We will utilize thematic analysis to identify and assess potential remaining barriers other than cost and access that inhibit the feasibility of pharmacogenetic testing in patients with medical complexity
Facilitators to acceptance of pharmacogenetic testing | 6 months
  Facilitators will be elicited through semi-structured interviews on consenting caregivers. We will utilize thematic analysis to identify and assess facilitators that enhance the feasibility of pharmacogenetic testing in patients with medical complexity

CONTACTS AND LOCATIONS:
Overall Officials: Sonya Tang Girdwood, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No specific Identifiable Patient Health Information (PHI) will be shared. However, aggregated data and de-identified info may be shared with IRB pre-approved collaborators.